CLINICAL TRIAL: NCT01482481
Title: Effectiveness of Implementing Nursing Care Plans Based on Scientific Methodology in Improving Metabolic and Blood Pressure Control of Type 2 Diabetes Mellitus Patients.
Brief Title: Effectiveness of Nursing Care Plans Based in Nursing Diagnoses in Metabolic Control of Type 2 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Hospital Carlos III, Madrid (Other)
Collaborators: Gerencia de Atención Primaria, Madrid (Other Government)
Responsible Party: Principal Investigator, Miguel Angel Salinero Fort, MD, Hospital Carlos III, Madrid
Other Study IDs: PI070865; 070865 (Other Grant/Funding Number: Instituto de la Salud Carlos III)
Record Dates: First submitted 2011-11-27; First posted 2011-11-30 (Estimated); Last update posted 2011-11-30 (Estimated); Status verified 2011-11

CONDITIONS: Type 2 Diabetes Mellitus; Cardiovascular Risk Factors
Keywords: Patient Care Planning; Type 2 Diabetes Mellitus; Cardiovascular Risk Factors; Primary Health Care; Spain
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Background: Nurses in clinical practice implement care to patients with Type 2 diabetes mellitus (DM2) in order to maintain normal blood glucose readings, promote weight loss and provide nutrition counseling to improve metabolic and blood pressure control. Because many disciplines contribute to patient's health outcomes, it is important to distinguish how nurses contribute to patient care and the achievement of health outcomes and the differences between the use or not the classification of Nursing Diagnoses, and the Nursing Interventions Classification (NIC) in clinical practice settings.

Methods: Prospective observational study with 2-year follow-up to assess the effect of Nursing Care Plans based on Scientific Methodology (NCPSM) on changing the control parameters in routine clinical practice conditions.

Settings: 31 Primary care centers in northeastern urban area of Madrid (Spain). Subjects: 24,124 DM2 patients (full universe).

DETAILED DESCRIPTION:
The computerized clinical record system (CCR) form for primary care of the Madrid Health Service was used as the data source. NCPSM was identified by clinical records of NANDA and NIC nursing taxonomies, and were defined as nursing care based on the following three criteria:

Criterion 1.- A patient's CCR must register valuation data based on Marjory Gordon "functional pattern" in at least the following areas:

* Health perception
* Nutritional-metabolic
* Activity-exercise. Criterion 2.- The problems identified and the proper management of treatment will be described using coded diagnoses with NANDA.

Criterion 3.- The nursing interventions carried out by standardized language will be registered according to the NIC taxonomy.

Eligibility criteria for patients were: older than 30 years of age, with previously diagnosed diabetes (cardinal clinical, plus random blood glucose >200 mg/dl or oral glucose of >200 mg/dl at 2 h, twice, or plasma fasting glucose of >126 mg/dl on two occasions or being diagnosed previously, received specific treatment for diabetes) and exclusion criteria were: gestational diabetes, patients involved in clinical trials, patients with life expectancy of less than one year (according to clinical judgment), homebound patients.

The primary outcome was HbA1c, lipid levels, blood pressure, and BMI after 24 and 48 months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* older than 30 years of age,
* with previously diagnosed diabetes (cardinal clinical, plus random blood glucose > 200 mg/dl or oral glucose of >200 mg/dl at 2 h, twice, or plasma fasting glucose of >126 mg/dl on two occasions or being diagnosed previously, received specific treatment for diabetes)

Exclusion Criteria:

* gestational diabetes,
* patients involved in clinical trials,
* patients with life expectancy of less than one year (according to clinical judgment),
* homebound patients

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 23,488 DM2 patients (full universe).
Sampling Method: Non-Probability Sample
Enrollment: 23488 (Actual)
Dates: Start 2008-01; Primary Completion 2009-12 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
HbA1c level | Final (before 4 years follow-up)

SECONDARY OUTCOMES:
Blood Pressure | Final (before 4 years follow-up)
Low-density lipoprotein (LDL) cholesterol | Final (before 4 years of follow-up)
Body Mass Index (BMI) | Final (before 4 years of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: JUAN CARDENAS, Study Director — Atención Primaria Madrid
Locations (1):
- Gerencia Atención Primaria, Madrid, Madrid, Spain

REFERENCES:
- [Derived] Cardenas-Valladolid J, Salinero-Fort MA, Gomez-Campelo P, de Burgos-Lunar C, Abanades-Herranz JC, Arnal-Selfa R, Andres AL. Effectiveness of standardized Nursing Care Plans in health outcomes in patients with type 2 Diabetes Mellitus: a two-year prospective follow-up study. PLoS One. 2012;7(8):e43870. doi: 10.1371/journal.pone.0043870. Epub 2012 Aug 27. PMID 22952794